CLINICAL TRIAL: NCT06938152
Title: Effects of Cycle Therapy With Romosozumab and Denosumab 2 Years vs 1 Year Romosozumab Followed by 1 Year Denosumab in Postmenopausal Osteoporosis Patients-A Randomized Control Trial
Brief Title: Effects of Cycle Therapy vs Sequential Therapy With Romosozumab and Denosumab in Postmenopausal Osteoporosis Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202501144MINE
Record Dates: First submitted 2025-04-06; First posted 2025-04-22 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-04

CONDITIONS: Osteoporosis; Osteoporosis Postmenopausal
Keywords: postmenopausal; Romosozumab; Denosumab; cycle therapy; Bone mineral density; Bone turnover marker
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal | interventions — romosozumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequential therapy group (Active Comparator): Romosozumab followed by Denosumab
  Interventions: Drug: Romosozumab followed by Denosumab
- Cycle therapy group (Experimental): Romosozumab and Denosumab Cycle Therapy
  Interventions: Drug: Romosozumab and Denosumab Cycle Therapy

INTERVENTIONS:
Drug: Romosozumab followed by Denosumab — Romosozumab 210mg/month for 12 months, then Denosumab 60mg/6months for 12 months
  Other Names: Sequential therapy group
  Arms: Sequential therapy group
Drug: Romosozumab and Denosumab Cycle Therapy — Romosozumab 210mg/month for 6 months then followed by Denosumab 60mg/6months once, and then repeat one more time after 6 months
  Other Names: Cycle therapy group
  Arms: Cycle therapy group

SUMMARY:
This study is a prospective, randomized, controlled clinical trial comparing the efficacy of a 24-month cyclic therapy regimen (6 months of Romosozumab followed by 6 months of Denosumab, repeated for two years) versus a traditional sequential treatment regimen (12 months of Romosozumab followed by 12 months of Denosumab). The goal is to determine which approach yields better therapeutic outcomes and to optimize drug strategies for osteoporosis patients.

DETAILED DESCRIPTION:
Osteoporosis is common in postmenopausal women and the elderly, and has been recognized by the World Health Organization as the second most prevalent metabolic bone disease worldwide. Most patients show no obvious symptoms, but a fall or sudden exertion can cause fragility fractures. Once fractures occur, complications such as acute pain, prolonged bed rest, and restricted mobility can significantly impact the quality of life and even increase mortality. Furthermore, managing these conditions requires substantial medical and social resources.

Currently, anti-osteoporosis medications are classified into two major categories: antiresorptive and anabolic agents. Studies have confirmed that both types can increase bone mineral density (BMD) and reduce fracture risk. However, each medication has usage limitations.

Denosumab is a potent antiresorptive drug, but long-term use can lead to rare side effects such as atypical femoral fractures (AFF) and medication-related osteonecrosis of the jaw (MRONJ). Additionally, stopping Denosumab can cause a severe rebound in bone resorption markers (CTX), leading to rapid BMD loss and an increased fracture risk. Managing drug discontinuation remains a major clinical challenge.

ELIGIBILITY:
Inclusion Criteria:

* 1. Postmenopausal women aged 50-90 years
* 2. BMD T-score ≤ -3.0 at any lumbar vertebra
* 3. Physically and mentally capable of understanding and complying with the study protocol and follow-up
* 4. Signed informed consent

Exclusion Criteria:

* 1. Previous osteoporosis treatment within the past two years, including Romosozumab, Teriparatide, Denosumab, Alendronate, Ibandronate, Zoledronic Acid, Risedronate, Raloxifene, or Bazedoxifene
* 2. Allergy to Romosozumab or Denosumab
* 3. Secondary osteoporosis
* 4. Autoimmune disease
* 5. Chronic steroid use (e.g., Chronic Obstruction Pulmonary Disease patients)
* 6. Hypercalcemia or hypocalcemia
* 7. Metabolic bone diseases
* 8. Primary or metastatic bone tumors
* 9. Cancer patients (except for in situ carcinoma and non-melanoma skin cancer, unless fully treated and in remission for five years)
* 10. Planned dental procedures (e.g., extractions, implants) within the next year
* 11. History of stent placement, myocardial infarction, stroke, or coronary artery disease
* 12. Renal disease (Creatinine > 1.5 mg/dL) or dialysis patients
* 13. Smoking more than one pack per day (except for those who have quit for over ten years)

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in bone mineral density (BMD) | Participants will undergo baseline assessments, followed by evaluations at 6, 12, 18 and 24 months.
  Change in BMD at lumbar spine, femoral neck and total hip at 24 months

SECONDARY OUTCOMES:
Change in bone turnover makers (BTM) level | Participants will undergo baseline assessments, followed by evaluations at 3, 6, 9, 12, 13, 15, 18, 21, and 24 months.
  Changes in BTM, including bone formation (P1NP) and resorption markers (CTX)
Change in visual Analogue Scale (VAS) score | Participants will undergo baseline assessments, followed by evaluations at 3, 6, 9, 12, 15, 18, 21, and 24 months.
  The Visual Analogue Scale (VAS) for pain will be used to assess participants' self-reported pain intensity. The VAS score ranges from 0 to 10, higher scores indicate worse pain intensity, and lower scores indicate less pain.
Oswestry Disability Index (ODI) score change | Participants will undergo baseline assessments, followed by evaluations at 6, 12, 18 and 24 months.
  The Oswestry Disability Index (ODI) will be used to assess the level of disability related to lower back pain. The ODI score ranges from 0 to 100, higher scores reflect worse functional disability and lower scores reflect better functional status.
New fracture | During the intervention period, up to 24 months.
  Any new fracture within 24 months
Adverse Events | During the intervention period, up to 24 months.
  Any adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kobayakawa T, Miyazaki A, Takahashi J, Nakamura Y. Verification of efficacy and safety of ibandronate or denosumab for postmenopausal osteoporosis after 12-month treatment with romosozumab as sequential therapy: The prospective VICTOR study. Bone. 2022 Sep;162:116480. doi: 10.1016/j.bone.2022.116480. Epub 2022 Jul 1. PMID 35787482
- [Result] Hong N, Shin S, Kim H, Cho SJ, Park JA, Rhee Y. Romosozumab following denosumab improves lumbar spine bone mineral density and trabecular bone score greater than denosumab continuation in postmenopausal women. J Bone Miner Res. 2025 Feb 2;40(2):184-192. doi: 10.1093/jbmr/zjae179. PMID 39485918
- [Result] Cosman F, Crittenden DB, Adachi JD, Binkley N, Czerwinski E, Ferrari S, Hofbauer LC, Lau E, Lewiecki EM, Miyauchi A, Zerbini CA, Milmont CE, Chen L, Maddox J, Meisner PD, Libanati C, Grauer A. Romosozumab Treatment in Postmenopausal Women with Osteoporosis. N Engl J Med. 2016 Oct 20;375(16):1532-1543. doi: 10.1056/NEJMoa1607948. Epub 2016 Sep 18. PMID 27641143
- [Result] Chandran M. The why and how of sequential and combination therapy in osteoporosis. A review of the current evidence. Arch Endocrinol Metab. 2022 Nov 11;66(5):724-738. doi: 10.20945/2359-3997000000564. PMID 36382762
- [Result] Gehrke B, Alves Coelho MC, Brasil d'Alva C, Madeira M. Long-term consequences of osteoporosis therapy with bisphosphonates. Arch Endocrinol Metab. 2023 Nov 10;68:e220334. doi: 10.20945/2359-4292-2022-0334. PMID 37948565
- [Result] McClung MR, Wagman RB, Miller PD, Wang A, Lewiecki EM. Observations following discontinuation of long-term denosumab therapy. Osteoporos Int. 2017 May;28(5):1723-1732. doi: 10.1007/s00198-017-3919-1. Epub 2017 Jan 31. PMID 28144701
- [Result] Cosman F, Huang S, McDermott M, Cummings SR. Multiple Vertebral Fractures After Denosumab Discontinuation: FREEDOM and FREEDOM Extension Trials Additional Post Hoc Analyses. J Bone Miner Res. 2022 Nov;37(11):2112-2120. doi: 10.1002/jbmr.4705. Epub 2022 Oct 12. PMID 36088628
- [Result] Reid IR, Billington EO. Drug therapy for osteoporosis in older adults. Lancet. 2022 Mar 12;399(10329):1080-1092. doi: 10.1016/S0140-6736(21)02646-5. PMID 35279261
- [Result] LeBoff MS, Greenspan SL, Insogna KL, Lewiecki EM, Saag KG, Singer AJ, Siris ES. The clinician's guide to prevention and treatment of osteoporosis. Osteoporos Int. 2022 Oct;33(10):2049-2102. doi: 10.1007/s00198-021-05900-y. Epub 2022 Apr 28. PMID 35478046
- [Result] Fogelman I, Blake GM. Different approaches to bone densitometry. J Nucl Med. 2000 Dec;41(12):2015-25. PMID 11138687
- [Result] Wang CY, Wu CH, Chen HM, Lin JW, Hsu CC, Chang YF, Tai TW, Fu SH, Hwang JS. Cost and effectiveness analyses of the anti-osteoporosis medication in patients with hip fracture in Taiwan: A population-based national claims database analysis. J Formos Med Assoc. 2023;122 Suppl 1:S92-S100. doi: 10.1016/j.jfma.2023.07.018. Epub 2023 Aug 11. PMID 37574339
- [Result] Wang CY, Fu SH, Yang RS, Shen LJ, Wu FL, Hsiao FY. Age- and gender-specific epidemiology, treatment patterns, and economic burden of osteoporosis and associated fracture in Taiwan between 2009 and 2013. Arch Osteoporos. 2017 Oct 25;12(1):92. doi: 10.1007/s11657-017-0385-5. PMID 29067572
- See also: National Institute of Arthritis and Musculoskeletal and Skin Diseases. (2022.12) — https://www.niams.nih.gov/health-topics/osteoporosis
- See also: 2023台灣成人骨質疏鬆防治之共識及指引 — https://www.toa1997.org.tw/download/files/2023台灣成人骨質疏鬆症防治之共識及指引_20230726_確認版(含封面).pdf